CLINICAL TRIAL: NCT06364930
Title: Sodium-glucose Co-transporter-2 Inhibitor (SGLT2i) to Prevent of Liver Complications in Patients With Chronic Hepatitis B and Diabetes Mellitus: a Double-blind, Randomised, Placebo-controlled Trial
Brief Title: SGLT2i to Prevent of Liver Complications in Patients With CHB and Diabetes Mellitus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGLT2i_HBV Study
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): 10mg QD for 60 months
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator): 10mg QD for 60 months
  Interventions: Drug: Placebo 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10mg Tab QD for 60 months.
  Arms: Dapagliflozin
Drug: Placebo 10mg Tab — Placebo 10mg Tab QD for 60 months.
  Arms: Placebo

SUMMARY:
This is a five-year, double blinded, randomised trial of dapagliflozin versus placebo in patients with chronic hepatitis B and DM or IFG complicated with compensated advanced chronic liver disease (cACLD). 412 subjects will be recruited. Subject will be randomly assigned to receive dapagliflozin 10mg daily or dapagliflozin placebo one tablet daily for up to 5 years. After randomization, subject will be followed up at month 3, month 6 and then 6-monthly until 60 months (follow up ± 4 weeks from scheduled clinic visit is allowed). At each visit, drug compliance, physical examination, observed or reported adverse events will be assessed. 10ml of blood will be taken at each visit and transient elastography to assess fibrosis regression will be performed at 60th month or at withdrawal visit. You are discouraged to use (pegylated)-interferon, any other NA including lamivudine, adefovir, and telbivudine, another SGLT2i Empagliflozin (Jardiance), Dapagliflozin + Metformin XR (Xigduo).

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection is a global health problem affecting approximately 234 million people worldwide; of those three-quarter come from the Asia-Pacific region.1 Up to 30%-40% of chronically infected persons will die of liver complications, including liver cancer and cirrhotic complications.2 The Global Burden of Disease Study 2016 revealed HBV as one of the top ten killers worldwide.3 Chronic HBV infection also represents a major global economic burden; with increasing socioeconomic costs.4 Majority of the liver complications and deaths is related to hepatocellular carcinoma (HCC) because of its high incidence rate and unfavourable clinical course.5

Sodium-glucose co-transporter-2 inhibitors (SGLT2i) is a potent antidiabetic agent that lowers blood glucose by inducing renal glycosuria.15 SGLT2i reduces cardiovascular and renal events by marked cardiac anti-fibrotic and anti-inflammatory effects,16 on top of dramatic weight reduction.6 A recent open-label, pilot study of nine patients with biopsy-proven non-alcoholic steatohepatitis (NASH) with type 2 DM received a SGLT2i (empagliflozin) 25 mg daily, for 24 weeks. SGLT2i led to histological improvement in steatosis, ballooning, and fibrosis, compared with historical placebo.7 SGLT2i also leads to more significant reduction of ALT.8 Several other randomised trials and cohort studies supported that SGLT2i also reduces liver fat content and liver fibrosis scores. SGLT2i has additional benefits on liver histology compared to other antidiabetic agents.8 The key pathways include control of hepatic inflammation and fibrosis, improvement of insulin resistance, and reduction of hepatic steatosis. The related mechanisms involve inflammatory parameters like high-sensitivity C-reactive protein, proinflammatory cytokines like interleukin-6 or TNF-alpha, reactive oxygen species and the inhibition of AMPc activation. The improvement was correlated with reductions in body weight, waist circumference and inflammatory parameters. The improvement was not correlated with changes in glucose control.9 All these favourable effects on liver have make it potentially useful to reduce liver complications.

Chronic hepatitis B is major cause of liver complications and death. Antiviral treatment with oral nucleos(t)ide analogues reduces but not abolish the risk of liver complications, especially in those with diabetes mellitus. Sodium-glucose co-transporter-2 inhibitors (SGLT2i) are promising in improving liver outcome in patients with chronic hepatitis B and diabetes mellitus. Our preliminary data provide strong plausibility that SGLT2i reduces the risk of liver complications. We are going to provide the definitive answer to this important clinical question through a randomised trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic hepatitis B on ETV, TDF or TAF monotherapy for at least 12 months.
2. Known or newly diagnosed type 2 diabetes mellitus (T2D), defined as HbA1c ≥5.7% or fasting blood sugar ≥5.6 mmol/L, or random blood sugar ≥11.1 mmol/L, or 2 hours sugar after oral glucose tolerance test ≥7.8 mmol/L.
3. Stable use of anti-diabetic drugs in the last three months.
4. Presence of compensated advanced chronic liver disease (cACLD) with liver stiffness measurement >10.0 kPa, or significant portal hypertension (spleen stiffness measurement > 41.3 kPa), or presence any sign of portal hypertension (e.g. splenomegaly, ascites, varices)
5. Aged 18 years old or above.
6. Written informed consent obtained.

Exclusion Criteria:

1. Patients with hepatitis C virus (HCV) infection as indicated by a positive antibody to HCV (anti-HCV) serology test.
2. Patients with history of cirrhotic complications or hepatocellular carcinoma
3. Patients with organ transplantation
4. Patients receiving a SGLT2i
5. Contraindications to SGLT2i due to renal insufficiency (GFR < 45 mL/min/1.73m2)
6. Poor glycaemic control with HbA1c >9.0%
7. Use of multiple anti-diabetic drugs (3 or more)
8. Change in anti-diabetic drugs in the last three months.
9. Serious medical illnesses or malignancy
10. Age < 18 years
11. No patient consents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is liver complications | 60 months
  defined as HCC and any cirrhotic complications, namely ascites, spontaneous bacterial peritonitis (SBP), variceal bleeding, hepatic encephalopathy, and/or hepatorenal syndrome (HRS).

SECONDARY OUTCOMES:
Cardiovascular complications | 60 months
  defined as cardiovascular deaths, hospitalizations for heart failure, and urgent heart failure
change in liver stiffness measurement | 60 months
  measured with transient elastography Unabbreviated scale title of kPa is kilopascals Minimum 0 kPa Maximum 80 kPa Higher scores mean a worse outcome
change anthropometric parameters (body weight) | 60 months
  body weight
change anthropometric parameters (waist-hip ratio) | 60 months
  waist-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Grace LH Wong, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarin SK, Kumar M, Eslam M, George J, Al Mahtab M, Akbar SMF, Jia J, Tian Q, Aggarwal R, Muljono DH, Omata M, Ooka Y, Han KH, Lee HW, Jafri W, Butt AS, Chong CH, Lim SG, Pwu RF, Chen DS. Liver diseases in the Asia-Pacific region: a Lancet Gastroenterology & Hepatology Commission. Lancet Gastroenterol Hepatol. 2020 Feb;5(2):167-228. doi: 10.1016/S2468-1253(19)30342-5. Epub 2019 Dec 15. PMID 31852635
- [Background] Likhitsup A, Lok AS. Understanding the Natural History of Hepatitis B Virus Infection and the New Definitions of Cure and the Endpoints of Clinical Trials. Clin Liver Dis. 2019 Aug;23(3):401-416. doi: 10.1016/j.cld.2019.04.002. Epub 2019 Jun 1. PMID 31266616
- [Background] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119
- [Background] Baik D, Kim BW, Oh JK, Kim KA, Ki M. Costs of viral hepatitis B in the Republic of Korea, 2002-2015. J Viral Hepat. 2020 Feb;27(2):156-167. doi: 10.1111/jvh.13219. Epub 2019 Nov 14. PMID 31638305
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Shrikrishnapalasuriyar N, Shaikh A, Ruslan AM, Sharaf G, Udiawar M, Price DE, Stephens JW. Dapagliflozin is associated with improved glycaemic control and weight reduction at 44 months of follow-up in a secondary care diabetes clinic in the UK. Diabetes Metab Syndr. 2020 May-Jun;14(3):237-239. doi: 10.1016/j.dsx.2020.03.007. Epub 2020 Mar 26. PMID 32247210
- [Background] Lai LL, Vethakkan SR, Nik Mustapha NR, Mahadeva S, Chan WK. Empagliflozin for the Treatment of Nonalcoholic Steatohepatitis in Patients with Type 2 Diabetes Mellitus. Dig Dis Sci. 2020 Feb;65(2):623-631. doi: 10.1007/s10620-019-5477-1. Epub 2019 Jan 25. PMID 30684076
- [Background] Leiter LA, Forst T, Polidori D, Balis DA, Xie J, Sha S. Effect of canagliflozin on liver function tests in patients with type 2 diabetes. Diabetes Metab. 2016 Feb;42(1):25-32. doi: 10.1016/j.diabet.2015.10.003. Epub 2015 Nov 11. PMID 26575250
- [Background] Carretero Gomez J, Ena J, Segui Ripoll JM, Carrasco-Sanchez FJ, Gomez Huelgas R, Casas Rojo JM, Suarez Tembra M, Carabantes Rueda JJ, Arevalo Lorido JC. Effect of newer antihyperglycemic drugs on liver steatosis indices in patients with diabetes and obesity. Curr Med Res Opin. 2021 Nov;37(11):1867-1873. doi: 10.1080/03007995.2021.1965563. Epub 2021 Aug 28. PMID 34357836
- [Background] Adamstein NH, Cornel JH, Davidson M, Libby P, de Remigis A, Jensen C, Ekstrom K, Ridker PM. Association of Interleukin 6 Inhibition With Ziltivekimab and the Neutrophil-Lymphocyte Ratio: A Secondary Analysis of the RESCUE Clinical Trial. JAMA Cardiol. 2023 Feb 1;8(2):177-181. doi: 10.1001/jamacardio.2022.4277. PMID 36449307